CLINICAL TRIAL: NCT01344733
Title: A Non - Interventional Study to Investigating the Ratio of Mis-diagnosed Bipolar Symptoms in Patient Diagnosed as With Treatment Resistant Major Depressive Disorder (MDD)
Brief Title: A Non Interventional Study to Investigating the Ratio of Mis-diagnosed Bipolar Symptoms in Patient With Major Depressive Disorder (MDD)
Acronym: Improve
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NIT-DUM-2010/1
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder; MDD
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDD: Patients with treatment resistant major depressive disorder will be evaluated in order to assess the presence of hypomanic symptoms as cause of resistance.

SUMMARY:
The study will only detect hypomanic symptoms in treatment resistant MDD patients by mean of HCL-32 administration. Further re-evaluation of MDD diagnosis is not a direct aim of the study. No efficacy and tolerability of pharmacological treatments will be assessed. Patients matching inclusion and exclusion criteria will be enrolled consecutively; each investigator will include the first 10 to 40 patients that will be visited as treatment resistant MDD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form
* Male and Female age: 18-65 years
* Diagnosis of MDD according to DSM-IV TR (296.3 x Major Depressive Disorder, recurrent)
* Treatment resistance defined as non-response to at least 2 antidepressants given in an ade

Exclusion Criteria:

* Patients already participating in clinical trial or any other interventional study
* Patients unable to understand HCL-32 item meaning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment resistant major depressive disorder will be evaluated in order to assess the presence of hypomanic symptoms as cause of resistance.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To define the potential bipolarity status in treatment resistant MDD patient population | 3 months
  assessment of presence of hypomanic symptoms, in order to reduce diagnostic mistakes leading to outcome worsening
Hypomanic condition will be defined if the patient will give positive answer to at least 12 items of HCL32. HCL-32-positive patients is expected to be ranged between 4.3% and 21.3%. The difference between the means in the two groups will be estimated. | 3 months

SECONDARY OUTCOMES:
To collect patient characteristics by evaluation of demographic information | 3 months
To collect disease characteristics by evaluation of the number of previous episodes, and the duration of current episode | 3 months
To collect information on the ongoing treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mauro Carta, Principal Investigator — A.O.U. Universitaria di Cagliari; Dr. Gino Montagnani, Study Chair — Astrazeneca Italy; Dr. Raffaele Sabia, Study Director — Astrazeneca Italy
Locations (29):
- Italy (29):
  - Research Site, Agrigento, AG
  - Research Site, Sciacca, AG
  - Research Site, Ancona, AN
  - Research Site, Corato, BA
  - Research Site, Putignano, BA
  - Research Site, Triggiano, BA
  - Research Site, Fasano, BR
  - Research Site, Bolzano, BZ
  - Research Site, Cagliari, CA
  - Research Site, Ortona, CH
  - Research Site, Cantù, CO
  - Research Site, Rogliano, CS
  - Research Site, Adrano-Bronte, CT
  - Research Site, Lamezia Terme, CZ
  - Research Site, Foggia, FG
  - Research Site, Firenze- ASL Di Firenze, FI
  - Research Site, Genova, GE
  - Research Site, Latina, LT
  - Research Site, Messina, ME
  - Research Site, Rho, MI
  - Research Site, Corleone, PA
  - Research Site, Palermo, PA
  - Research Site, Guidonia, RM
  - Research Site, Roma, RM
  - Research Site, Capaccio, SA
  - Research Site, Savona, SA
  - Research Site, Montecchio Maggiore, VI
  - Research Site, Castellammare di Stabia
  - Research Site, Novara